CLINICAL TRIAL: NCT04267263
Title: A Novel Approach to Reducing Adiposity Among Young Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM20015458
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Weight Loss; Men; Lifestyle Risk Reduction; Cardiovascular Diseases; Obesity
MeSH Terms: conditions — Weight Loss; Multiple Endocrine Neoplasia Type 1; Risk Reduction Behavior; Cardiovascular Diseases; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed Treatment Control group (No Intervention): Participants will receive the treatment after completion of the 3-month follow-up assessment
- Lifestyle group (Experimental): Participants will receive the treatment immediately
  Interventions: Behavioral: Self-guided lifestyle intervention

INTERVENTIONS:
Behavioral: Self-guided lifestyle intervention — The intervention will consist of one 60-minute group based online session, adapted specifically for young men based previous work with young adults, followed by a self-guided program for 12-weeks. Participants will receive a tool kit that includes evidence-based resources (scale for self-weighing, handouts that will include free self-monitoring apps and strategies for no-cost exercise, sample meal plans and meal planning tips, and tips for healthy living that emphasize risk areas) to assist them during the self-guided phase, as well as weekly health risk text messages.
  Arms: Lifestyle group

SUMMARY:
The purpose of this research study is to find out whether a primarily self-guided program can produce changes in weight, body fat and cardiovascular risk among young men.

DETAILED DESCRIPTION:
This self-guided lifestyle intervention may help men to reduce weight and improve heart health because it has been adapted to meet the possible weight loss needs of young men. Young men may experience reductions in body weight after enrollment in the intervention, but this is unknown.

Study participation lasts approximately 3 months. Participants will be assessed by the study staff and fill out questionnaires about current lifestyle practices (diet, physical activity, sleep habits, risk behaviors). Weight, medical events, and medication use within the last 3 months will be assessed. Eligible participants will be randomly assigned (like the flip of a coin) to the control group or self-guided group.

ELIGIBILITY:
Inclusion Criteria:

1. self-identify as a man
2. 18-35 years old
3. BMI 25-45kg/m2
4. Live in North America

Exclusion Criteria:

1. an uncontrolled medical condition that might make it unsafe to change their eating or engage in unsupervised physical activity (e.g., uncontrolled hypertension)
2. a diagnosis of Type 1 or Type 2 diabetes
3. report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q), which will be administered during prescreen
4. currently enrolled in another weight loss program, taking weight loss medication or history of weight loss surgery
5. change in medication(s) within the last 3 months that could influence weight (e.g., steroids)
6. have lost > 5% body weight within the last 3 months
7. report a history of anorexia nervosa or bulimia nervosa or any compensatory behaviors within the previous 3 months
8. report hospitalization for a psychiatric condition within the last year
9. report high alcohol intake (AUDIT score > 16).
10. are not able to speak and read English
11. do not possess a mobile device or are unwilling to use it to receive study text messages
12. Given strict data regulations outside of North America (i.e., Europe), we will only include participants living in North America (i.e., United States, Canada).

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Self-identified males
Enrollment: 35 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Percent weight lost | 3 months
  Percent weight change (measured in kg via calibrated scale); calculated as: (post-treatment weight - baseline weight) / baseline weight *100

SECONDARY OUTCOMES:
Change in perceived risk for heart disease | Baseline to 3 months
  Perceived risk assessed via 12-item Risk Behavior Diagnosis scale
Change in minutes of moderate to vigorous physical activity | Baseline to 3 months
  Physical activity assessed via 21-item Global Physical Activity Questionnaire
Change in diet quality | Baseline to 3 months
  Dietary habits assessed via 26-item National Cancer Institute's Dietary Screening Questionnaire
Change in sleep quality | Baseline to 3 months
  Sleep habits assessed via 6-item Common Elements Sleep Quesitonnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jessica G LaRose, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University School of Medicine, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reading JM, Crane MM, Guan J, Jackman R, Thomson MD, LaRose JG. Acceptability of a Self-Guided Lifestyle Intervention Among Young Men: Mixed Methods Analysis of Pilot Findings. JMIR Form Res. 2024 Apr 5;8:e53841. doi: 10.2196/53841. PMID 38578686
- [Derived] Reading JM, Crane MM, Carlyle K, Perera RA, LaRose JG. A Self-Guided Lifestyle Intervention for Young Men: Findings from the ACTIVATE Randomized Pilot Trial. J Mens Health. 2022;18(9):191. doi: 10.31083/j.jomh1809191. Epub 2022 Sep 14. PMID 36846742

DOCUMENTS (1):
  • Informed Consent Form (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT04267263/ICF_000.pdf